CLINICAL TRIAL: NCT02232113
Title: The Response of Continuous Erythropoietic Receptor Activator (CERA) With Different Dose Interval and the Survey for Influence Factors
Brief Title: Frequent Dosing of CERA Improves Nutrition and Inflammation in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Chih-Ching Lin,M.D PhD., Taipei Veterans General Hospital, Taiwan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-10-004IA
Record Dates: First submitted 2014-08-03; First posted 2014-09-05 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Anemia; Inflammation; Malnutrition
Keywords: malnutrition, inflammation, and anemia (MIA) syndrome,; hemodialysis,; erythropoietin stimulating agent (ESA),; cost-effectiveness,; pharmacokinetics,; endothelial dysfunction
MeSH Terms: conditions — Anemia; Inflammation; Malnutrition; Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CERA (Experimental): We included HD patients with stable hematocrit (between 30~36%) under intravenous administration of CERA 100 μg once monthly for two months. Then they were shifted to receive CERA 50μg twice monthly for anther two months and finally they were shifted back to receive CERA 100 μg once monthly again for additional two months. Then we compared the hematocrit, nutrition status and inflammation markers every two months for 6 months totally. Those who had bleeding or received surgery or blood transfusion were excluded.
  Interventions: Drug: CERA

INTERVENTIONS:
Drug: CERA — changing frequency of administration from once to twice monthly under a fixed total monthly dose of CERA
  Other Names: Full name: Continuous Erythropoietic Receptor Activator; Abbreviation : CERA; Generic name: Methoxy polyethylene glycol-epoetin beta; Brand name：Mircera®

SUMMARY:
The response of Continuous Erythropoietic Receptor Activator (CERA) with different dose interval and the survey for influence factors:

We aim to evaluate a better clinical response which can be achieved by different dosing interval of a fixed dose of CERA. We expect this study can determine the dosing schedule with better clinical response to CERA and identify the associated factors predicting the cost-effectiveness of CERA in maintenance hemodialysis (HD) patients in Taiwan.

DETAILED DESCRIPTION:
We included HD patients with stable hematocrit (between 30~36%) under intravenous administration of CERA 100 μg once monthly for two months. Then they were shifted to receive CERA 50μg twice monthly for anther two months and finally they were shifted back to receive CERA 100 μg once monthly again for additional two months. Then we measured and compared the erythropoietic response (hematocrit, hemoglobin), profiles of iron status as well as nutritional status and inflammatory markers among the study subjects every two months for a total of 6 months. Those who had bleeding or received surgery or blood transfusion were excluded.

ELIGIBILITY:
Inclusion Criteria:

* HD patients with stable hematocrit (between 30~36%) under intravenous administration of CERA 100 μg once monthly for two months.

Exclusion Criteria:

* HD patients were excluded due to active bleeding (major trauma, gastric ulcer bleeding, or surgery), blood transfusion or administration of additional erythropoietic stimulating agent (ESA) other than CERA within the follow-up period during the study perod of 6 months. People who discontinued CERA as their ESA were also excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2012-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Erythropoietic response | every 2 months for six months
  We measured and compared the hematocrit, hemoglobin, and iron status profiles (ferritin, iron, total iron binding capacity) among those enrolled patients every 2 months for 6 months totally.

SECONDARY OUTCOMES:
Nutritional status and inflammatory markers | every 2 months for a total of 6 months
  Nutritional status (albumin, prealbumin) and inflammatory markers [interleukin 6, tumor necrosis factor-α (TNF-α)]

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Ching Lin, MD, PhD, Study Director — Division of Nephrology and Department of Medicine, Taipei Veterans General Hospital
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Liu WS, Wu YL, Li SY, Yang WC, Chen TW, Lin CC. The waveform fluctuation and the clinical factors of the initial and sustained erythropoietic response to continuous erythropoietin receptor activator in hemodialysis patients. ScientificWorldJournal. 2012;2012:157437. doi: 10.1100/2012/157437. Epub 2012 Apr 19. PMID 22619601
- See also: Used to treat patients with symptomatic anaemia associated with chronic kidney disease (CKD). — http://www.roche.com/products/product-details.htm?type=product&id=83